CLINICAL TRIAL: NCT03230435
Title: Health Related Quality of Life for Patients With Anorexia Nervosa in Denmark.
Acronym: QOLAN-DK
Status: Active, not recruiting | Type: Observational
Sponsor: René Klinkby Støving (Other)
Collaborators: Region of Southern Denmark (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, René Klinkby Støving, Professor, PhD, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: QOLAN-DK 10226757
Record Dates: First submitted 2017-07-20; First posted 2017-07-26 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Anorexia Nervosa; Health-Related Quality Of Life
Keywords: anorexia nervosa, health-related quality of life
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anorexia nervosa: Treatment settings as usual.
  Interventions: Other: Treatment settings as usual.
- Healthy controls: No interventions.

INTERVENTIONS:
Other: Treatment settings as usual. — Treatment according to guidelines and the local instructions (psychotherapy and dietary guidance).
  Groups: Anorexia nervosa

SUMMARY:
Eating disorders (ED) comprise a multitude of symptoms involving a disturbed body image and a preoccupation with food or bodyweight. EDs are often difficult to treat, in part due to the lack of motivation for improvement. Anorexia nervosa (AN) has the highest mortality rate of any psychiatric disease, and less than half of patients will recover from the disease. Studies have found that patients suffering from AN have impaired health-related quality of life (HRQoL) compared to the general population. It has also been suggested that despite improvement in clinical parameters, patients report deterioration in HRQoL, which is in line with a study finding low agreement between patient perceived outcome and clinician assessed characteristics. To evaluate the patients' perception of their disease, it is important to develop reliable and valid assessment tools. Previously generic questionnaires have been used to assess HRQoL in Danish ED patients, as no disease-specific questionnaires have been developed. Translating and validating a disease-specific questionnaire would provide a useful tool in assessing current treatment and in developing new treatment options. This study aimed to develop a Danish version of an internationally disease-specific HRQoL questionnaire. Furthermore, HRQoL is assessed in patients who have gone through shorter or longer treatment.

DETAILED DESCRIPTION:
INTRODUCTION Anorexia nervosa (AN) is an eating disorder of unknown etiology. The evidence base for treatment is still very limited considering the extent to which this disorder erodes lives and still carries the highest fatality rate of any psychiatric disease as well as any other chronic disease in adolescence.

There is no consensus on appropriate effect goals in AN. Assessment of biomedical parameters alone is not sufficient, why evaluation tools that consider the patient's own perception of their health and well-being are essential. However, patients with AN characteristically have a different opinion of their needs to that of the health professionals, which can lead to differences in treatment goals, ambivalence towards treatment, and immense compliance difficulties.

Health-related quality of life (HRQOL) can be defined as the overall effect of a medical condition and/or its consequent therapy upon a patient. HRQOL is subjective and multidimensional, encompassing physical and occupational function, psychological state, social interaction and somatic sensation. Discrepancy between one's current level of function and one's ideals or expectations can result in lower self-rated HRQOL, while cognitive flexibility is believed to contribute to good HRQOL. Patients with AN typically have unrealistically high expectations of themselves, are often rigid and usually do not consider weight gain to be a necessity for a positive outcome. Therefore, treatment may potentially lead to further reduction of HRQOL (for example due to coerced hospitalization), despite significant positive improvements in biomedical parameters.

In a recently published meta-analysis examining the HRQOL of patients with eating disorders, several methodological challenges were identified such as variations in study design, diagnostic criteria and health outcome measurement. It is essential that HRQOL measures are valid and reliable for the patient group in question. These measures can be either generic (applicable to all patient groups) or disease-specific (designed to detect HRQOL changes specific to a disease).

Only a few disease-specific HRQOL measures for AN have been developed. The Eating Disorder Quality of Life (EDQLS) questionnaire was published by a Canadian research group and consists of 40 items on selected topics including relationships with family and others, physical and psychological health and eating. Subsequent studies have shown that the EDQLS demonstrates excellent psychometric properties in terms of validity, reliability and responsiveness to change.

OBJECTIVES

1. To validate a Danish version of the Eating Disorder Quality of Life questionnaire in two age ranges, 13-17 years and +18 years in patients with AN.
2. To assess age-specific HRQoL in patients with AN in different treatment settings.

DESIGN Preparatory study: Testing and adaptation of the Danish version of the EDQLS for use by 13-17 year olds with anorexia nervosa.

Study 1: Concurrent validity and internal consistency. EDQLS, ED symptomatology, distress, social function and generic HRQOL assessed in different clinical samples of AN patients aged 13-17 & +18 years and in a sample of age-matched healthy controls within a normal weight range.

Study 2: Test-retest reliability. EDQLS completed twice with a 2-4-week interval in a sample of weight- and treatment-stable outpatients and controls aged 13-17 & +18 years.

Study 3: Sensitivity to change. EDQLS applied three times over a 4-6-week interval in a sample of AN inpatients aged 13-17 & +18 years.

Study 4: Patients outside the established treatment. EDQLS, ED symptomatology, distress, social function and generic HRQoL score among members and followers with BMI<18 recruited from the official website for the national patient organizations.

METHODS

TRANSLATION Prior to this study, the initial translations of the EDQLS was carried out using the method recommended by WHO World Mental Health Initiative Translation Guidelines. After permission from the Canadian authors, an expert panel of bilingual staff from an ED outpatient clinic worked on the translation from English to Danish, aiming for conceptual equivalence between the versions (i.e. similar relevance and meaning in the two languages/cultures). After panel discussions to create a consensus version the Danish draft questionnaire was completed individually by 18 adult women with AN, who in subsequent qualitative interviews commented on their understanding of the items and any difficulties they had with the wording. The linguistic comments and suggestions from the patients were used to further improve the translation, which was then approved by the expert panel. This draft was back-translated and the back-translation was reviewed by the Canadian authors of the scale. After the refinement of a single word, it was accepted as the official Danish EDQLS translation. Both the Danish version and the original EDQLS are licensed.

In the present study, the original EDQLS will be tested and adjusted as necessary for use patients aged 13-17 years. This will be done by repeating the qualitative interviews with six adolescents AN patients (13-17 years) to investigate whether the questionnaire should be linguistically modified for this age group. Any modifications will be discussed with the Canadian developers of EDQLS.

MEASURES Screening questionnaire: Patients will be asked to fill out a questionnaire regarding current weight, height and information regarding current medication.

Disease-specific quality of life (EDQLS). WHO-5 Well-being Index (WHO-5). Generic health related quality of life: Short Form-36 (SF-36). Eating disorder symptomatology: Eating Disorder Inventory-3. Depression: The Beck Depression Inventory II (BDI-II). Impairment in functioning: Work and Social Adjustment Scale (WSAS). Total item burden: Total amount of measures is 201 items. Estimated time for administration is about two hours. The questionnaires are stored in RedCap, automatically uploading the answers as the patients fill them out.

DATA ANALYSES AND STATISTICS

POWER CALCULATIONS The sample size is based on the validation work of the original language version in Canada. A high response rate of at least 80% is expected because there is a high participatory interest in the subject and purpose of the study, and because the participants receive a small fee.

MULTIVARIATE ANALYSES Description of the subsamples is presented as means and standard deviations and frequencies. Inter-item correlations and confirmatory factor analyses are performed on the full sample across age-groups and health status and in sub-populations. Pearson correlations are produced for the included symptom and HRQOL scores.

ETHICAL CONSIDERATIONS According to Danish legislation, surveys are exempt from ethical board review. However, a formal enquiry was made and the ethical board determined that the project was approved without further application to the ethical committee. Participants will be informed that study participation is voluntary, and will have no effect on their treatment and management. There are no risks associated with participating in the study.

All questionnaires and tests used in the study are validated, recommended and widely distributed clinically for diagnosing in psychiatry.

To facilitate a high proportion of completion, all participants (patients and controls) who complete the test are honored with Danish kroner (DDK) 150.

ANONYMITY The project is approved by the Data Protection Agency, File no. 17/3218. The data will be stored in a data sheet, REDCap.

FINANCE The study is a 100 % non-commercial study. The Jascha Fund has supported the post doc salary for 18 months. There will be applied for licenses, participation fees, and operating expenses.

DISSEMINATION AND TENTATIVE PUBLICATIONS

The study findings, both positive and negative results, will be disseminated through communication at congresses and written scientific publications. Publications will be made according to the Vancouver criteria with the tentative titles:

* Health-related quality of life in anorexia nervosa: Validation of a Danish language version in young and adult patients.
* In-patients treatment of anorexia nervosa: Does it improve health related quality of life?
* Patients with anorexia nervosa, not seeking established treatment: specific health related quality of life.
* Gender differences in health-related quality of life in patients with anorexia nervosa.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients fulfilling Diagnostic and Statistical Manual of Mental Disorders, version 5 (DSM-5) criteria for anorexia nervosa.

EXCLUSION CRITERIA

1. Patients and controls who are unable to complete a Danish language questionnaire.
2. Controls: Any medication, except vitamins or oral contraceptives.

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — 90-95% female can be expected among patients with AN. The controls are matched on gender.
Study Population: PATIENTS will be recruited through specialized centres in Denmark and through contact to Patient Association's network.
  CONTROLS will be identified through public call for proposals. The proposals will be posted at institutions of further education and public schools in Odense with students in the appropriate age range.
Sampling Method: Probability Sample
Enrollment: 496 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
EDQLS | through a hospitalization, an average of 5 weeks
  Disease specific health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: René K Støving, PhD, Principal Investigator — Center for Eating Disorders, Odense University Hospital, & Psychiatric survived in Southern Denmark
Locations (1):
- Department of Endocrinology, Center for Eating Disorders, Odense UH, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data will be stored at Odense patient Data Explorative Network (OPEN).

REFERENCES:
- [Background] Winkler LA, Frolich JS, Gudex C, Horder K, Bilenberg N, Stoving RK. Patient- and clinician- reported outcome in eating disorders. Psychiatry Res. 2017 Jan;247:230-235. doi: 10.1016/j.psychres.2016.11.047. Epub 2016 Nov 30. PMID 27923148
- [Background] Winkler LA, Christiansen E, Lichtenstein MB, Hansen NB, Bilenberg N, Stoving RK. Quality of life in eating disorders: a meta-analysis. Psychiatry Res. 2014 Sep 30;219(1):1-9. doi: 10.1016/j.psychres.2014.05.002. Epub 2014 May 14. PMID 24857566
- [Background] Winkler LA, Bilenberg N, Horder K, Stoving RK. Does specialization of treatment influence mortality in eating disorders?--A comparison of two retrospective cohorts. Psychiatry Res. 2015 Dec 15;230(2):165-71. doi: 10.1016/j.psychres.2015.08.032. Epub 2015 Aug 28. PMID 26391650
- [Background] Adair CE, Marcoux GC, Cram BS, Ewashen CJ, Chafe J, Cassin SE, Pinzon J, Gusella JL, Geller J, Scattolon Y, Fergusson P, Styles L, Brown KE. Development and multi-site validation of a new condition-specific quality of life measure for eating disorders. Health Qual Life Outcomes. 2007 Apr 30;5:23. doi: 10.1186/1477-7525-5-23. PMID 17470290
- [Background] Adair CE, Marcoux GC, Bischoff TF, Cram BS, Ewashen CJ, Pinzon J, Gusella JL, Geller J, Scattolon Y, Fergusson P, Styles L, Brown KE. Responsiveness of the Eating Disorders Quality of Life Scale (EDQLS) in a longitudinal multi-site sample. Health Qual Life Outcomes. 2010 Aug 11;8:83. doi: 10.1186/1477-7525-8-83. PMID 20701776
- [Background] Winkler LA, Hemmingsen SD, Gudex C, Blegvad AC, Stoving RK, Arnfred SMH. A Danish translation of the eating disorder quality of life scale (EDQLS). J Eat Disord. 2019 May 1;7:11. doi: 10.1186/s40337-019-0241-7. eCollection 2019. PMID 31069077